CLINICAL TRIAL: NCT00980642
Title: Accuracy of the Draeger Dual-sensor Temperature Measurement System in The Perioperative Period
Brief Title: Accuracy of the Drager Dual-sensor Temperature Measurement System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrea Kurz, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08-453
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Hypothermia; Anesthesia
Keywords: surgery; thermometer; non-invasive; interoperative core temperature; anesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia (Other): Temperature is measured by Draeger double-sensor and esophageal stethoscope temperature sensor every 5-min during the surgery.
  Interventions: Device: Draeger double-sensor; Device: Esophageal stethoscope temperature sensor
- Regional anesthesia (Other): Temperature is measured by Draeger double-sensor and Foley catheter temperature sensor every 5-min during the surgery.
  Interventions: Device: Draeger double-sensor; Device: Foley catheter temperature sensor

INTERVENTIONS:
Device: Draeger double-sensor — The sensor will be attached to the patient's forehead with adhesive tape, and a small amount of contact gel will be applied between sensor and skin.
Device: Esophageal stethoscope temperature sensor — Esophageal temperature is measured by sensors incorporated into an esophageal stethoscope during the surgery.
  Arms: General anesthesia
Device: Foley catheter temperature sensor — Urinary bladder temperature is measured via a sensor incorporated into a Foley catheter during the surgery
  Arms: Regional anesthesia

SUMMARY:
Our primary hypothesis is that the Draeger dual-sensor temperature monitoring system, used at the forehead, is sufficiently accurate compared to tympanic, bladder or esophageal temperature and oral temperature for routine clinical use during hypothermic conditions, as well as during fever.

DETAILED DESCRIPTION:
We will include patients undergoing general anesthesia or regional anesthesia. The temperature recorded by Draeger dual-sensor monitoring system will be obtained at 5-minute interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing trauma surgery with general anesthesia
* Patients undergoing orthopedic surgery with regional anesthesia

Exclusion Criteria:

* Younger than 18 or older than 80 years of age
* Have a pre-existing nasogastric tube
* Require bispectral index monitoring
* Upper esophageal disease
* Forehead rash or infection
* Oral infection or trauma
* Ear infection or drainage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, M.D., Principal Investigator — The Cleveland Clinic; Daniel I Sessler, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients having trauma surgery with general anesthesia were recruited from the University of Vienna, while patients having orthopedic surgery with regional anesthesia were recruited from the Cleveland Clinic from January 2009 to June 2011.
Period: Overall Study
Arm/Group | General Anesthesia | Regional Anesthesia
Started | 36 | 20
Completed | 36 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia | Regional Anesthesia | Total
Number analyzed (Participants) | 36 | 20 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [19 to 80] | 65 [47 to 79] | 64 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 14 | 7 | 21
Region of Enrollment [Number; unit: participants]
  United States | 0 | 20 | 20
  Austria | 36 | 0 | 36
Ambient temperature [Mean (Standard Deviation); unit: Celsius degree] | 19.2 (1.2) | 19.5 (1.0) | 19.4 (1.1)
Duration of surgery [Median (Inter-Quartile Range); unit: hours] | 2.0 [1.1 to 3.0] | 1.2 [0.7 to 1.5] | 1.8 [1.0 to 2.2]

OUTCOME MEASURES:

1. Primary Outcome: The Bias Between Temperature Measured by Drager Double-sensor vs Core Temperature
Description: Determine if the Drager double-sensor temperature monitoring system, used at the forehead is accurate compared to esophageal temperature for general anesthesia group and bladder temperature for regional anesthesia group.
Time Frame: From anesthesia induction to the end of surgery
Measure: Mean (95% Confidence Interval); unit: Celsius degree
Arm/Group | General Anesthesia | Regional Anesthesia
Number analyzed (Participants) | 36 | 20
Celsius degree | -0.01 [-0.61 to 0.59] | -0.13 [-0.65 to 0.40]

2. Secondary Outcome: Sensitivity for Detection of Hypothermia
Description: Hypothermia is defined as a temperature < 36 Celsius degree
Time Frame: From anesthesia induction to the end of surgery
Measure: Number (95% Confidence Interval); unit: percent of hypothermias
Arm/Group | General Anesthesia | Regional Anesthesia
Number analyzed (Participants) | 36 | 20
percent of hypothermias | 0.70 [0.48 to 1.00] | 0.83 [0.68 to 1.00]

3. Secondary Outcome: Specificity for Detection of Hypothermia
Description: Hypothermia will be defined as a temperature < 36 Celsius degree
Time Frame: From anesthesia induction to the end of surgery
Measure: Number (95% Confidence Interval); unit: percent of non-hypothermias
Arm/Group | General Anesthesia | Regional Anesthesia
Number analyzed (Participants) | 36 | 20
percent of non-hypothermias | 0.78 [0.68 to 0.95] | 0.69 [0.34 to 1.00]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 3 hours
Arm/Group | General Anesthesia | Regional Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/20
Other Adverse Events (participants affected / at risk) | 0/36 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes